CLINICAL TRIAL: NCT04067986
Title: Camrelizumab Combined With Apatinib in the Treatment of Patients With Advanced Gastric Cancer and Colorectal Cancer：One-arm Exploratory Clinical Trial
Brief Title: Camrelizumab Combined With Apatinib in the Treatment of Patients With Advanced Gastric Cancer and Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Arise-FJ-R301
Record Dates: First submitted 2019-08-14; First posted 2019-08-28 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Colorectal Cancer Recurrent
MeSH Terms: interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab + Apatinib (Other): Camrelizumab + Apatinib
  Interventions: Drug: Camrelizumab; Drug: Apatinib

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab One course will last 28 days.Intravenous injection at a dose of 200 mg, q2w
  One course will last 28 days. Oral administration at a dose of 250 mg/d
  Other Names: Apatinib
Drug: Apatinib — Apatinib One course will last 28 days.Oral administration at a dose of 250 mg, qd

SUMMARY:
The efficacy and safety of the use of Camrelizumab combined with Apatinib

DETAILED DESCRIPTION:
To evaluate the clinical efficacy and safety of Camrelizumab combined with Apatinib in the treatment of patients with advanced gastric cancer and colorectal cancer.

The 62 patients were enrolled in a 2-week regimen with 200mg Camrelizumab given intravenously every two weeks and 250mg apatinib mesylate every 4 weeks for a treatment cycle until progressive or intolerable，then the objective remission rate(ORR) was calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years；
* Patients with histologically or cytologically confirmed advanced or metastatic gastric cancer and colorectal cancer.
* Patients who had previously progressed after receiving standard second-line advanced treatment；
* Patients with at least one evaluable or measurable lesions as per RECIST version 1.1 （CT scan length and diameter of tumor lesion≥10mm，CT scan of lymph node lesion was short diameter≥15mm，scan slice thickness 5mm；）
* ECOG performance status (PS) 0 - 2；
* Life expectancy of at least 3 months；
* Patients with adequate organ function at the time of enrollment as defined below:

  1. Blood routine examination standard：（without blood transfusion within 14 days before enrollment）

     1. Hb ≥90g/L，
     2. WBC≥3.0×109/L
     3. ANC ≥ 1.5×109/L，
     4. PLT ≥ 80×109/L；
  2. Biochemical examination shall meet the following standards：

     1. BIL <1.5 times the upper limit of normal（ULN），
     2. ALT and aspartate aminotransferase (AST) <2.5×upper limit of normal (ULN)，If liver metastasis is present，ALT and AST<5ULN ；
     3. Serum creatinine Cr≤1ULN，Serum creatinine >50ml/min（Cockcroft-Gault math）
* Women of childbearing age in the serum or urine pregnancy test is negative within 7 days prior to study enrollment and must be Non-lactating patients，and agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 8 months after the end of the study； males should agree to patients who must use contraception during the study period and within 8 months after the end of the study period
* Subjects voluntarily joined the study, signed informed consent, good compliance, and followed up;

Exclusion Criteria:

* Except for other malignant tumors, basal cell carcinoma of the skin and cervical cancer in situ in the past 5 years；
* Patients who have undergone systemic chemotherapy, radiotherapy, surgery, hormone therapy, or immunotherapy <2 weeks before enrollment；
* With severe heart, liver, lung and kidney disease；Significant neurological or psychiatric disorders；Patients with partial or complete gastrointestinal obstruction；
* Patients with a large amount of pleural effusion or ascites requiring drainage；
* Patients with symptomatic brain metastasis；
* Patients with hypertension that is difficult to control (systolic blood pressure ≥140 mmHg and diastolic blood pressure ≥90 mmHg) despite treatment with several hypotensive agents; Patients with acute coronary syndrome (including myocardial infarction and unstable angina), and with a history of coronary angioplasty or stent placement performed within 6 months before enrollment；Patients with acute coronary syndrome（included QTc male>450ms，female>470ms）and cardiac dysfunction；
* Women who are pregnant or breastfeeding；
* Patients with concurrent autoimmune disease, or a history of chronic or recurrent autoimmune disease;
* Patients with concurrent autoimmune disease, or a history of chronic or recurrent autoimmune disease: included HIV positive or a history of organ transplantation and allogeneic bone marrow transplantation;
* Patients with interstitial lung disease with symptoms or signs of activity；
* Patients with a risk of gastrointestinal bleeding may not be enrolled, including the following: (1) active digestive ulcer lesions and fecal occult blood (++); (2) nausea and hematemesis within 2 months Medical history. Simple fecal occult blood (+) is not an exclusion criterion；Coagulation abnormalities （INR>1.5、APTT>1.5ULN）；
* Urine protein ≥ ++ or confirmed 24 hour urine protein quantitation；
* Patients with non-healing wound, non-healing ulcer, or non-healing bone fracture;
* Patients with a seizure disorder who require pharmacotherapy；
* Patients with a history of hypersensitivity to any of the study drugs, similar drugs, or excipients；
* The investigator believes that there are any conditions that may damage the subject or result in the subject being unable to meet or perform the research request;
* participated in other clinical studies before and during treatment；

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-09-23 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | one year
  Objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumours (RECIST) version. 1.1, and immune-related (ir) RECIST

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse-Events | one year
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Li Xiao, Doctor, Principal Investigator — Zhongshan Hospital Xiamen University
Locations (1):
- Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No